CLINICAL TRIAL: NCT01809808
Title: A Prospective Study of Outcome After Therapy for Acromegaly
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine, Columbia University
Other Study IDs: AAAA0890; R56DK064720 (NIH)
Record Dates: First submitted 2012-08-08; First posted 2013-03-13 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Acromegaly
Keywords: Acromegaly; Pituitary tumor
MeSH Terms: conditions — Acromegaly; Pituitary Neoplasms | interventions — Surgical Procedures, Operative; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acromegaly Subjects: People who have a biochemical diagnosis of acromegaly, and will or have already undergone surgery for acromegaly and will be taking medications for acromegaly . Subjects will undergo blood sampling, metabolic rate measurement, adipose tissue biopsy and total body magnetic resonance imaging before and over time after either surgery or medical therapy for acromegaly.
  Interventions: Procedure: Surgery for acromegaly; Drug: Medications for acromegaly; Diagnostic Test: Total body magnetic resonance imaging; Procedure: Adipose Tissue Biopsy
- Healthy Subjects: People who are not diagnosed with acromegaly, responding to flyer or by word of mouth for participation, without medical problems, not taking medications, and with a stable weight for 3 months prior to study. Subjects will undergo blood sampling, total body MRI and adipose tissue biopsy once.
  Interventions: Diagnostic Test: Total body magnetic resonance imaging; Procedure: Adipose Tissue Biopsy

INTERVENTIONS:
Procedure: Surgery for acromegaly — (non-experimental) standard procedure
  Groups: Acromegaly Subjects
Drug: Medications for acromegaly — (non-experimental) standard procedure
  Other Names: Drugs used to lower growth hormone
  Groups: Acromegaly Subjects
Diagnostic Test: Total body magnetic resonance imaging — Subjects will undergo total body MRI with spectroscopy of the muscle and liver before and 3-6 months, 12 and 24 months after surgery or medical therapy for acromegaly.
Procedure: Adipose Tissue Biopsy — Subjects will undergo biopsy of subcutaneous adipose tissue before and 12 and 24 months after surgery or medical therapy for acromegaly.

SUMMARY:
The purpose of this study is to evaluate hormone values and other markers of disease activity in a cohort of patients with acromegaly at the time of diagnosis and then prospectively after surgical or other treatment. This study is designed to determine blood levels of growth hormone and related hormones and cardiovascular risk markers as well as signs and symptoms of the disease at diagnosis and how these parameters change over time after surgical or other therapy. The investigators will also obtain hormonal data in a group of 50 healthy subjects who will each be studied just once with an oral glucose tolerance test (OGTT). These data will provide a comparison group to the acromegaly subjects.

DETAILED DESCRIPTION:
Surgical removal of the pituitary tumor is the usual first form of treatment offered, but this is curative in only approximately 70% of patients. If not adequately treated, the disease can have significant morbidity largely due to the development of hypertension, diabetes and malignancy as well as possible loss of vision or other neurologic complications of a large pituitary mass. Inadequately treated acromegaly is also associated with a mortality rate 2-3 fold over the general population. All the mechanisms responsible for the increased morbidity and mortality in acromegaly as well as what biochemical criteria should be used during treatment in order to normalize the increased morbidity and mortality are not known. This study aims to follow patients with acromegaly prospectively from active disease through treatment in order to identify these factors.

ELIGIBILITY:
Acromegaly Subjects

Inclusion Criteria:

* Adult males and females.
* Ages 18 and over.
* Presenting to the PI or one of the sub-investigators for evaluation of acromegaly.
* Must have a biochemical diagnosis of acromegaly consisting of an elevated serum insulin-like growth factor 1 (IGF-1) level. Supportive although not required for entry are an elevated growth hormone (GH) level and a failure of GH to suppress normally after oral glucose administration.
* Willingness to participate in this study's procedures.

Exclusion Criteria:

* Subjects who are unwilling to comply with the procedures outlined in the study.
* Subjects who do not have the ability to fully comprehend the nature of the study, to follow instructions, and/or cooperate with study procedures
* Are unwilling to provide informed consent to participate in the study.

Healthy Subjects

Inclusion Criteria:

* Adult males and females.
* Ages 18 and over.
* Responding to ads for participation or by word of mount.
* No medical problems, no medications, stable weight for 3 months prior to study.
* Willingness to participate in this study's procedures.

Exclusion Criteria:

* Subjects who are unwilling to comply with the procedures outlined in the study.
* Subjects who do not have the ability to fully comprehend the nature of the study, to follow instructions, and/or cooperate with study procedures
* Are unwilling to provide informed consent to participate in the study.
* Failure to meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects newly diagnosed with acromegaly or who have previously undergone surgery for acromegaly are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2025-08 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
Biochemical activity of Acromegaly | At 5 years after therapy for acromegaly
  The study will assess the status of biochemical disease activity of acromegaly before and after treatment for acromegaly. Blood samples are taken for fasting growth hormone and insulin-like growth factor 1 and growth hormone levels 60, 90 and 120 minutes after oral glucose taken at baseline visit, post-operative or after the initiation of medical therapy at month 1 (fasting blood only), month 3 (fasting blood only), month 6, month 12, and annual assessments for at least 5 years.

SECONDARY OUTCOMES:
Visceral Adipose Tissue Mass | Before therapy, 6 months, 1 year and 2 years after the intervention, surgery or medical therapy.
  Total Body Magnetic Resonance Imaging
Intra-hepatic Lipid | Before therapy, 6 months, 1 year and 2 years after the intervention, surgery or medical therapy.
  Proton magnetic resonance spectroscopy of liver
Resting metabolic rate | Before, 1 year and 2 years after the intervention
  Measurement of resting metabolic rate by indirect calorimetry
Intra-myocellular lipid | Before therapy, 6 months, 1 year and 2 years after the intervention, surgery or medical therapy.
  Proton magnetic resonance spectroscopy of soleus muscle
Relative expression of CD11c gene | Before, 1 year and 2 years after the intervention
  Relative expression of CD11c gene in biopsied subcutaneous adipose tissue
Relative expression of CD68 gene | Before, 1 year and 2 years after the intervention
  Relative expression of CD68 gene in biopsied subcutaneous adipose tissue
Relative expression of MCP1 gene | Before, 1 year and 2 years after the intervention
  Relative expression of MCP1 gene in biopsied subcutaneous adipose tissue
Relative expression of IL6 gene | Before, 1 year and 2 years after the intervention
  Relative expression of IL6 gene in biopsied subcutaneous adipose tissue
Plasma levels of c-reactive protein | Before, 1 year and 2 years after the intervention
  Levels of c-reactive protein in peripheral venous blood
Plasma Levels of ghrelin | Before, 1 month, 3 months, 6 months, 1 year and 2 years after intervention
  Levels of ghrelin in peripheral blood
Plasma Levels of AgRP | Before, 1 month, 3 months, 6 months, 1 year and 2 years after intervention
  Levels of AgRP in peripheral blood
Plasma Levels of GLP1 | Before, 1 month, 3 months, 6 months, 1 year and 2 years after intervention
  Levels of GLP1 in peripheral blood
Serum Levels of insulin | Before, 1 month, 3 months, 6 months, 1 year and 2 years after intervention
  Levels of insulin in peripheral blood
Serum Levels of glucose | Before, 1 month, 3 months, 6 months, 1 year and 2 years after intervention
  Levels of glucose in peripheral blood
Serum Levels of glucagon | Before, 1 month, 3 months, 6 months, 1 year and 2 years after intervention
  Levels of glucagon in peripheral blood
Serum Levels of GIP | Before, 1 month, 3 months, 6 months, 1 year and 2 years after intervention
  Levels of GIP in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U Freda, M.D., Principal Investigator — Columbia University
Locations (1):
- Neuroendocrine Unit; Columbia University Medical Center, 180 Fort Washington Avenue 9-970, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freda PU, Reyes-Vidal C, Jin Z, Pugh M, Panigrahi SK, Bruce JN, Wardlaw SL. Plasma Agouti-Related Protein Levels in Acromegaly and Effects of Surgical or Pegvisomant Therapy. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5453-5461. doi: 10.1210/jc.2019-01079. PMID 31361303
- [Derived] Reyes-Vidal CM, Mojahed H, Shen W, Jin Z, Arias-Mendoza F, Fernandez JC, Gallagher D, Bruce JN, Post KD, Freda PU. Adipose Tissue Redistribution and Ectopic Lipid Deposition in Active Acromegaly and Effects of Surgical Treatment. J Clin Endocrinol Metab. 2015 Aug;100(8):2946-55. doi: 10.1210/jc.2015-1917. Epub 2015 Jun 2. PMID 26037515
- [Derived] Reyes-Vidal C, Fernandez JC, Bruce JN, Crisman C, Conwell IM, Kostadinov J, Geer EB, Post KD, Freda PU. Prospective study of surgical treatment of acromegaly: effects on ghrelin, weight, adiposity, and markers of CV risk. J Clin Endocrinol Metab. 2014 Nov;99(11):4124-32. doi: 10.1210/jc.2014-2259. Epub 2014 Aug 19. PMID 25137427
- See also: Columbia University Medical Center: Neuroendocrine Diseases Program — https://www.columbiaendocrinology.com/neuroendocrine